CLINICAL TRIAL: NCT00509483
Title: Long-Term Follow-up and Outcome of Administering Recombinant Human Thyrotropin as an Adjuvant of Therapy With Radioiodine in the Outpatient Treatment of Multinodular Goitres
Brief Title: Three-Year Follow-up of Radioiodine Therapy for Goitre
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRN 833/02
Record Dates: First submitted 2007-07-27; First posted 2007-07-31 (Estimated); Last update posted 2008-10-17 (Estimated); Status verified 2008-10

CONDITIONS: Tratment of Multinodular Goitre
Keywords: multinodular; goitre; recombinant human TSH
MeSH Terms: conditions — Goiter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: Radioactive iodine — Radioactive iodine preceded by rhTSH

SUMMARY:
Background: Preadministration of recombinant human thyrotropin (rhTSH) increases the amount and homogeneity of thyroid radioiodine uptake, and when used as an adjuvant can augment the efficiency of 131I therapy by allowing multinodular goitre (MNG) volume reduction.

Objective: The investigators aimed to assess low-dose rhTSH-aided fixed-activity radioiodine therapy outcome in MNG patients.

Design: This was a long-term (36 months) observational study. Methods: The investigators measured 24 h thyroid radioiodine uptake (RAIU) of 1.4 µCi (0.5 MBq) of 131-iodine at baseline and 24 h after intramuscular injection of 0.1 mg rhTSH in 42 patients (aged 42-80 years) who subsequently received 30 mCi 131-iodine 24 h after an identical rhTSH injection. Urinary iodine was measured at baseline and at 3 months after following a low iodine diet. TSH, free thyroxine (FT4), T3 (T3) and thyroglobulin (TG) were measured at baseline, 24 h, 48 h, 72 h, 168 h, one month, 3, 6, 9, 12, 18, 24 and 36 months after therapy. Thyroid volume was assessed by computer tomography at baseline and every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients with multinodular goitre

Exclusion Criteria:

* Aversion to any form of treatment
* Previous radioiodine therapy
* Being unable to complete a prolonged follow-up; and
* Having serious cardiovascular disorders.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2002-01; Study Completion 2006-12

CONTACTS AND LOCATIONS:
Overall Officials: Rossana Romão, MD, Principal Investigator — University of Sao Paulo